CLINICAL TRIAL: NCT05631743
Title: A Virtual Reality-assisted Cognitive Behavior Therapy With Inuit in Quebec - a Proof-of-concept Randomized Controlled Trial
Brief Title: VR-CBT With Inuit in Quebec
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); MedTeq (Industry); Douglas Foundation (Unknown); McGill University (Other)
Responsible Party: Principal Investigator, Martin Lepage, James McGill professor, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUSMD 21-52
Record Dates: First submitted 2022-10-21; First posted 2022-11-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Emotion Regulation
Keywords: virtual reality; cognitive behavioural therapy
MeSH Terms: conditions — Emotional Regulation | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: The study design is a proof-of-concept, two-arm RCT with a VR-assisted therapist -guided psychotherapy and self-management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR-CBT (Experimental): A trained psychotherapist provides CBT-VR for up to 10 sessions over 10 weeks.
  Interventions: Behavioral: VR-CBT
- Self-management (Active Comparator): Participants use a commercial VR application at home for guided self-management at their own pace over 10 weeks.
  Interventions: Behavioral: Self-management

INTERVENTIONS:
Behavioral: VR-CBT — The therapy is focused on emotion regulation through guided learning in virtual reality. The manual is a modified conventional cognitive behavioral therapy to include these aspects and the suggestions of an advisory committee of Inuit and non-Inuit health service providers (e.g., cultural adaptation).
  Arms: VR-CBT
Behavioral: Self-management — The previously developed commercial VR program involves guided relaxation and meditation techniques.
  Arms: Self-management

SUMMARY:
The study design is a two-arm randomized controlled pilot trial. The investigators will recruit Inuit in Montreal and randomly assign them to two treatment groups (n=20 each). The active psychotherapy group will receive a ten-week manualized virtual reality (VR) assisted cognitive-behavioral psychotherapy (VR-CBT) at the clinic and guided by a psychotherapist. The VR-CBT will aim at improving emotion regulation. The comparison group will use a VR self-management program, Calm Place, for guided relaxation during ten weeks at home. To evaluate outcome in both groups, the researchers will measure self-reports of emotion regulation, affect, distress and well-being, as well as a psychophysiological reactivity paradigm pre-post treatment.

DETAILED DESCRIPTION:
In this protocol, the investigators present a proof-of-concept trial that will evaluate an active psychotherapy and self-management, both targeting emotion regulation skills. The study design is a two-arm randomized controlled trial. The investigators will recruit Inuit and randomly assign them to two treatment groups (n=20 each). The active psychotherapy group will receive a ten-week manualized virtual reality (VR) assisted cognitive-behavioral psychotherapy (VR-CBT) at the clinic and guided by a psychotherapist. The VR-CBT will aim at improving emotion regulation, a set of skills or competence that is impacted by traumatic experiences and mediates the effect of trauma on psychiatric symptoms. The investigators conducted a cultural adaptation of the therapy for Inuit with a co-design grounded in qualitative participatory methods. The comparison group will use a VR self-management program, Calm Place, for guided relaxation during ten weeks at home. To evaluate outcome in both groups, the researchers will include a psychophysiological reactivity paradigm pre-post treatment and self-reports of emotion regulation, anxiety, mood, substance use, functionality and quality of life. The investigators expect to see preliminary evidence that our VR-CBT can be more successful than guided VR relaxation with Calm Place (self-management) decreasing difficulties in emotion regulation, psychiatry symptoms, increasing well-being, and normalizing responses to stressful stimuli (reactivity).

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as Inuk
2. Live in Montreal
3. be between 14 to 60 years of age
4. be proficient in English or French
5. No history of cardiac conditions
6. No history of epilepsy
7. Can provide an emergency contact
8. Tolerance of VR headset
9. Tolerance of sensors
10. Has no current suicidal or homicidal risk
11. No history of psychosis or schizophrenia
12. Current stable mood
13. Is generally mentally stable
14. Score less than 8 on the Alcohol Use Disorders Identification Test C
15. Score less than 3 on the Drug Abuse Screen Test (10 item version)
16. Not have had any change in psychoactive medications during 4 weeks preceding screening and inclusion to the study

Exclusion Criteria:

1. does not identify as Inuk
2. youth below the age of 14 and adults above the age of 60.
3. self-reported history of psychosis or schizophrenia
4. current substance abuse, as measured by two screens (AUDIT-C, DAST-10)
5. other mental or physical condition that might preclude them from the trial (i.e., pre-existing heart conditions, convulsions, acute mental health risk).

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation | Approximately 5 minutes
  Difficulties in Emotion Regulation Scale-16 is a short, valid measure of emotion regulation, scored from 16(low difficulties)-80 (higher difficulties).

SECONDARY OUTCOMES:
heart rate | Approximately 1 hour testing session.
  The participants undergo a psychophysiological reactivity testing paradigm, where we measure heart rate (in beats per minute) during a baseline, forest walk and height exposure in VR. The paradigm testing will be done during the initial visit and the last visit after the end of the VR intervention (minimum of seven and maximum of ten weeks). We measure changes in reactivity and resting level responses as compared from relaxed (forest walk) to height exposure, expecting lower resting levels of heart rate.
heart rate variability | Approximately 1 hour testing session.
  The participants undergo a psychophysiological reactivity testing paradigm, where we measure heart rate variability baseline, forest walk and height exposure in VR. The paradigm testing will be done during the initial visit and the last visit after the end of the VR intervention (minimum of seven and maximum of ten weeks). We measure changes in reactivity as compared from relaxed (forest walk) to height exposure, increased heart rate variability.
skin conductance response | Approximately 1 hour testing session.
  The participants undergo a psychophysiological reactivity testing paradigm, where we measure skin conductance during a baseline, forest walk and height exposure in VR. The paradigm testing will be done during the initial visit and the last visit after the end of the VR intervention (minimum of seven and maximum of ten weeks). We measure changes in reactivity and resting level responses as compared from relaxed (forest walk) to height exposure, expecting decreased skin conductance response.
anxiety (momentary) | Approximately 1 hour testing session.
  The participants undergo a psychophysiological reactivity testing paradigm, involving during a baseline, forest walk and height exposure in VR. The paradigm testing will be done during the initial visit and the last visit after the end of the VR intervention (minimum of seven and maximum of ten weeks). Visual analogue scales for anxiety are given during each segment of this test, scored 0 to 100 (not at all anxious- very anxious).
emotional arousal (momentary) | Approximately 1 hour testing session.
  The participants undergo a psychophysiological reactivity testing paradigm, involving during a baseline, forest walk and height exposure in VR. The paradigm testing will be done during the initial visit and the last visit after the end of the VR intervention (minimum of seven and maximum of ten weeks). Visual analogue scales for emotional arousal are given during each segment of this test, scored 0-100 (very calm- very excited).
emotional valence (momentary) | Approximately 1 hour testing session.
  The participants undergo a psychophysiological reactivity testing paradigm, involving during a baseline, forest walk and height exposure in VR. The paradigm testing will be done during the initial visit and the last visit after the end of the VR intervention (minimum of seven and maximum of ten weeks). Visual analogue scales for emotional valence are given during each segment of this test, scored 0-100 (very pleasant-very unpleasant).
Psychiatric Symptoms (anxiety) | Administration time is around 3 minutes
  We will monitor any change in psychiatric symptom severity, and any loss/gain of probable psychiatric diagnosis (for screening measures), expecting severity of symptoms to decrease. Generalized Anxiety Disorder Scale-7 is a scale scored 0-21 (minimal anxiety to severe anxiety).
Psychiatric Symptoms (depression) | Administration time is around 4 minutes
  We will monitor any change in psychiatric symptom severity, and any loss/gain of probable psychiatric diagnosis (for screening measures), expecting severity of symptoms to decrease. Patient Health Questionnaire - 9 is a scale scored 0-27 (minimal to severe).
Psychiatric Symptoms (post traumatic stress disorder) | Administration time is between 2 minutes
  We will monitor any change in psychiatric symptom severity, and any loss/gain of probable psychiatric diagnosis (for screening measures), expecting severity of symptoms to decrease. Primary Care Screen for Post-Traumatic Stress Disorder for Diagnostic and Statistical Manual-5 (PC-PTSD-5) is a screening, measure where a score of 3 indicates probable post-traumatic stress.
Psychiatric Symptoms (alcohol use disorder) | Administration time is between 2 minutes
  We will monitor any change in psychiatric symptom severity, and any loss/gain of probable psychiatric diagnosis (for screening measures), expecting severity of symptoms to decrease. Alcohol Use Disorders Identification Test- C screens for probably alcohol use disorder with a score of 3 or 4.
Psychiatric Symptoms (substance use disorders) | Administration time is between 4 minutes
  We will monitor any change in psychiatric symptom severity, and any loss/gain of probable psychiatric diagnosis (for screening measures), expecting severity of symptoms to decrease. Drug Abuse Screening Test-10 is a scale scored from 0-10, with higher scores indicating more intensive assessment needed.
Psychological distress and well being: Clinical outcome in routine evaluation outcome measure and 10 item (CORE- OM/10) | Approximately 10 minutes
  We will monitor any change in psychological well-being, as measured by a scale for psychological distress (constituted by multiple subscales including well being). The scale can operate as a screening tool with a score of 10 or 11.
Psychological distress and well being: Short/ Warwick Edinburgh Mental Wellbeing Scale | Approximately 10 minutes
  We will monitor any change in psychological well-being, as measured by a scale which covers mental wellbeing as a feeling and function, expecting wellbeing to increase and distress to decrease. Higher scores indicate higher wellbeing (short version is scored 7-35; long version 14-70).
Feasibility of interventions (attendance/useage) | 10 weeks of intervention period (researcher recorded)
  The number (percentages) of sessions attended (or completed at home) will serve as indicators of feasibility.
Feasibility of interventions (treatment completion) | 10 weeks of intervention period (researcher recorded)
  Treatment completion (minimum of 7 sessions of VR in either arm) and drop-outs will serve as indicators of feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Outi Linnaranta, MD, Ph.D, Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada